CLINICAL TRIAL: NCT07390370
Title: Establishment of a Registry for Immediate Drug Allergy
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2025-1428
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Drug Hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Collect whole blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immediate drug hypersensitivity reactions are acute adverse reactions that occur within one hour of drug administration and can result in life-threatening symptoms such as urticaria, angioedema, and anaphylaxis. Current diagnostic methods have high false-negative and false-positive rates, and standardized testing for non-IgE-mediated reactions (e.g., MRGPRX2) is lacking. This creates significant gaps in patient safety and clinical decision-making.

The study aims to establish a registry of patients with immediate drug hypersensitivity reactions to analyze clinical characteristics and investigate the underlying mechanisms of IgE-mediated and non-IgE-mediated reactions. Blood samples will be collected prospectively, using residual serum from routine clinical tests where available, to minimize additional blood draws. Mechanistic analyses will focus on IgE-mediated and non-IgE-mediated pathways, including MRGPRX2 expression in mast cells and basophils, and measurement of active β-tryptase as a biomarker for anaphylaxis.

In addition, a retrospective review will be conducted of medical records from the last 10 years to identify causative drugs and classify the underlying mechanisms of hypersensitivity. Based on this, specific target drugs will be selected for further prospective analysis. Data and biospecimens from participants in an existing allergy registry, who consent to secondary use, will also be included in the study.

Through the integration of clinical data and multi-layered biomarker analysis, the study aims to improve understanding of immediate drug hypersensitivity mechanisms and develop predictive models. Ultimately, this research will contribute to the establishment of personalized diagnosis, prevention, and treatment strategies for drug allergies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 19 years or older diagnosed with immediate hypersensitivity reactions (such as rash, urticaria, angioedema, anaphylaxis, etc.) within 1 hour after drug administration."
2. Utilization of samples and clinical data from patients with immediate drug hypersensitivity who consented to participate in secondary research, registered in the study 'Establishment of a Registry for Identifying Factors Related to Diagnosis, Treatment, and Prognosis in Allergic Disease Patients' (Project Number 4-2013-0397).

Exclusion Criteria:

1. Participants who do not consent to participate in the study."
2. Children and adolescents under the age of 19."
3. Participants who are unable to read or understand the consent form."

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 19 years or older diagnosed with immediate hypersensitivity reactions (such as rash, urticaria, angioedema, anaphylaxis, etc.) within 1 hour after drug administration.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Endotype Classification and Basophil Activation in Immediate Drug Hypersensitivity | 4 years
  Derivation and classification of endotype clusters in immediate drug hypersensitivity reactions based on basophil/mast cell activation markers and mediator-release profiles.

SECONDARY OUTCOMES:
Biomarker Associations with Endotypes and Clinical Phenotypes in Drug Hypersensitivity | 4 years
  1. Association of MRGPRX2-related markers with endotype clusters and clinical phenotypes in immediate drug hypersensitivity reactions.
  2. Association of serum β-tryptase with endotype clusters and anaphylaxis/severity phenotypes.
  3. Exploratory identification of candidate biomarkers from stool and/or skin specimens associated with endotype clusters.

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share individual participant data (IPD) from this registry study with qualified researchers conducting non-commercial research. The shared data will include clinical data, laboratory test results, and biological samples (e.g., blood, stool). Data sharing will be subject to the following conditions:
  1. Researchers must submit a formal request detailing the proposed research and data use.
  2. Data will be de-identified to protect confidentiality and ensure ethical compliance.
  3. Data is for non-commercial use only and cannot be used commercially without prior consent.
  4. Recipients must obtain ethics or IRB approval.
  5. Data will be shared via a secure platform, and recipients must sign a data use agreement (DUA).
  6. Access will be provided for 5 years post-study, after which data will be archived or deleted.